CLINICAL TRIAL: NCT06527885
Title: Treatment Satisfaction and Effectiveness of Lurasidone on Quality of Life and Functioning in Adult Patients With Schizophrenia Treated in the Real World Italian Clinical Practice
Brief Title: Lurasidone Non-Interventional Study in Schizophrenia Patients
Status: Completed | Type: Observational
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Other Study IDs: 153(A)IM21322
Record Dates: First submitted 2024-07-26; First posted 2024-07-30 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Schizophrenia
Keywords: Lurasidone; Patient's treatment satisfaction; Quality of Life; Functioning changes; Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Lurasidone Treatment: Adult patients suffering from schizophrenia treated for 3 months with lurasidone according to routine clinical practice.
  Interventions: Drug: Lurasidone

INTERVENTIONS:
Drug: Lurasidone — Patients treated with Lurasidone in according to routine clinical practice, in Italy

SUMMARY:
The study is a multicentric, national, non-interventional, prospective, single arm study.

The main goal of this study is to gather information about the effects, in a real-life setting, of lurasidone treatment on patient's reported outcomes, in terms of patient's treatment satisfaction, Quality of Life and functioning changes after 6 weeks from lurasidone treatment initiation in schizophrenia patients naïve to lurasidone.

DETAILED DESCRIPTION:
Important aim of the study is to investigate, aspects related to effectiveness, safety and tolerability at 3 months' lurasidone treatment in a routine practice in Italian clinical settings.

Only patients with primary diagnosis of schizophrenia who are prescribed lurasidone was evaluated for inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years) male or female subjects;
* Primary diagnosis of schizophrenia
* Patients not previously treated with lurasidone. The choice to initiate lurasidone treatment is independent of being included in the study;
* Patients legally capable of giving their written consent for participation in the study and for personal data processing.

Exclusion Criteria:

* Concomitant participation in a clinical trial

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from schizophrenia treated with lurasidone, according to routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Patient's and caregiver's treatment satisfaction- releif of symptoms | 6 weeks after treatment
  Patient's and caregiver's satisfaction is evaluated by Seven-point Likert scales derived from Treatment Satisfaction Questionnaire for Medication used to assess patient's and caregiver's satisfaction about efficacy, safety, usability and global impression of medications.
  Patient's satisfaction with efficacy, safety, ease of use, and overall impression of medication was measured using seven-point Likert scales derived from the Treatment Satisfaction Questionnaire for Medication. Caregiver's satisfaction with efficacy, safety, ease of use, and overall impact on patient management was assessed using seven-point Likert scales derived from the Treatment Satisfaction Questionnaire for Medication. The questionnaire consists of 4 items. Each item is scored on a 7-point Likert scale ranging from 1 (Extremely dissatisfied) to 7 (Extremely satisfied).
Patient's functioning & quality of life | 6 weeks after treatment
  To assess the Patient's functioning and quality of life a Quality-of-Life Scale was used.
  Quality Life Scale is a standardized questionnaire that evaluates various aspects of an individual's life, interpersonal relation, instrumental role, Intrapsychic Foundations, Common Objects and Activities and overall satisfaction with life.
  The Quality of Life Scale is a validated measure of health-related quality of life and functioning in schizophrenia that focuses on intrapsychic, social, and negative symptoms and their impact on functioning in schizophrenia. The questionnaire consists of 21 items in 4 domains: Interpersonal Relations (8 items), Instrumental Role (4 items), Intrapsychic Foundations (7 items), and Common Objects and Activities (2 items). Each item is scored on a 7-point Likert scale ranging from 0 (severe impairment) to 6 (normal or unimpaired functioning). A score is calculated for each domain, and the total score ranges from 0 to 126.

SECONDARY OUTCOMES:
Patient's and caregiver's treatment satisfaction- releif of symptoms | 3 months after treatment
  Patient's and caregiver's satisfaction was evaluated by Seven-point Likert scales derived from Treatment Satisfaction Questionnaire for Medication used to assess patient's and caregiver's satisfaction about efficacy, safety, usability and global impression of medications.
  Patient's satisfaction with efficacy, safety, ease of use, and overall impression of medication was measured using seven-point Likert scales derived from the Treatment Satisfaction Questionnaire for Medication. Caregiver's satisfaction with efficacy, safety, ease of use, and overall impact on patient management was assessed using seven-point Likert scales derived from the Treatment Satisfaction Questionnaire for Medication. The questionnaire consists of 4 items. Each item is scored on a 7-point Likert scale ranging from 1 (Extremely dissatisfied) to 7 (Extremely satisfied).
Patient's functioning & quality of life | 3 months after treatment
  To assess the Patient's functioning and quality of life a Quality-of-Life Scale was used.
  Quality Life Scale is a standardized questionnaire that evaluates various aspects of an individual's life, interpersonal relation, instrumental role, Intrapsychic Foundations, Common Objects and Activities and overall satisfaction with life.
  The Quality of Life Scale is a validated measure of health-related quality of life and functioning in schizophrenia that focuses on intrapsychic, social, and negative symptoms and their impact on functioning in schizophrenia. The questionnaire consists of 21 items in 4 domains: Interpersonal Relations (8 items), Instrumental Role (4 items), Intrapsychic Foundations (7 items), and Common Objects and Activities (2 items). Each item is scored on a 7-point Likert scale ranging from 0 (severe impairment) to 6 (normal or unimpaired functioning). A score is calculated for each domain, and the total score ranges from 0 to 126.
Evaluation of adverse drug reactions, akathisia, other extrapyramidal symptoms by Investigator's Assessment Questionnaire | 3 months after treatment
  To assess the safety a Investigator's Assessment Questionnaire was used. Investigator's Assessment Questionnaire is a validated, clinician-rated scale, designed to assess relative effectiveness (efficacy, safety, and tolerability) of antipsychotic medications in patients with schizophrenia. The Investigator's Assessment Questionnaire consists of 12 equally weighted items: positive symptoms, negative symptoms, other efficacy symptoms, somnolence, weight gain, signs and symptoms of prolactin elevation, akathisia, other extrapyramidal symptoms, other safety or tolerability issues, cognition, energy, and mood. For each item, the current medication was compared with previous antipsychotic medication on a five-point scale from 1 (much better) to 5 (much worse). Total Investigator's Assessment Questionnaire scores range from 12 to 60 with lower Investigator's Assessment Questionnaire total scores indicating better relative treatment effectiveness.
Evaluation of the weight gain, signs and symptoms of prolactinby by Investigator's Assessment Questionnaire | 3 months after treatment
  To assess the tolerability a Investigator's Assessment Questionnaire was used. Investigator's Assessment Questionnaire is a validated, clinician-rated scale, designed to assess relative effectiveness (efficacy, safety, and tolerability) of antipsychotic medications in patients with schizophrenia. The Investigator's Assessment Questionnaire consists of 12 equally weighted items: positive symptoms, negative symptoms, other efficacy symptoms, somnolence, weight gain, signs and symptoms of prolactin elevation, akathisia, other extrapyramidal symptoms, other safety or tolerability issues, cognition, energy, and mood. For each item, the current medication was compared with previous antipsychotic medication on a five-point scale from 1 (much better) to 5 (much worse). Total Investigator's Assessment Questionnaire scores range from 12 to 60 with lower Investigator's Assessment Questionnaire total scores indicating better relative treatment effectiveness.
Efficacy evaluation by Clinical global impression | 6 weeks after treatment
  To assess the efficacy a Clinical Global Impression - Severity of Illness is used.
  Clinical Global Impression - Severity of Illness measures the clinician's impression of the patient's current state of mental illness on a 7-point scale ranging from 1 (normal-not at all ill) to 7 (among the most extremely ill patients). Although Clinical Global Impression - Severity is considered a very simple and synthetic tool to assess the severity of schizophrenia it has been demonstrated that it is nonetheless reliable and its indications were consistent with other more sophisticated scales such as Global Assessment of Functioning and Positive and Negative Syndrome Scale . The Clinical Global Impression - Severity requires the knowledge of the patient's clinical history; for this reason, the patient should always be assessed by the same physician in order to detect any change in the patient's condition.
Efficacy evaluation by Clinical global impression | 3 months after treatment
  To assess the efficacy a Clinical Global Impression - Severity of Illness is used.
  Clinical Global Impression - Severity of Illness measures the clinician's impression of the patient's current state of mental illness on a 7-point scale ranging from 1 (normal-not at all ill) to 7 (among the most extremely ill patients). Although Clinical Global Impression - Severity is considered a very simple and synthetic tool to assess the severity of schizophrenia it has been demonstrated that it is nonetheless reliable and its indications were consistent with other more sophisticated scales such as Global Assessment of Functioning and Positive and Negative Syndrome Scale. The Clinical Global Impression - Severity requires the knowledge of the patient's clinical history; for this reason, the patient should always be assessed by the same physician in order to detect any change in the patient's condition.
Efficacy evaluation by Investigator's Assessment Questionnaire | 6 weeks after treatment
  To assess the efficacy a Investigator's Assessment Questionnaire is used.
  Investigator's Assessment Questionnaire is a validated, clinician-rated scale, designed to assess relative effectiveness (efficacy, safety, and tolerability) of antipsychotic medications in patients with schizophrenia. The Investigator's Assessment Questionnaire consists of 12 equally weighted items: positive symptoms, negative symptoms, other efficacy symptoms, somnolence, weight gain, signs and symptoms of prolactin elevation, akathisia, other extrapyramidal symptoms, other safety or tolerability issues, cognition, energy, and mood. For each item, the current medication was compared with previous antipsychotic medication on a five-point scale from 1 (much better) to 5 (much worse). Total Investigator's Assessment Questionnaire scores range from 12 to 60 with lower Investigator's Assessment Questionnaire total scores indicating better relative treatment effectiveness.
Efficacy evaluation by Investigator's Assessment Questionnaire | 3 months after treament
  To assess the efficacy a Investigator's Assessment Questionnaire is used.
  Investigator's Assessment Questionnaire is a validated, clinician-rated scale, designed to assess relative effectiveness (efficacy, safety, and tolerability) of antipsychotic medications in patients with schizophrenia. The Investigator's Assessment Questionnaire consists of 12 equally weighted items: positive symptoms, negative symptoms, other efficacy symptoms, somnolence, weight gain, signs and symptoms of prolactin elevation, akathisia, other extrapyramidal symptoms, other safety or tolerability issues, cognition, energy, and mood. For each item, the current medication was compared with previous antipsychotic medication on a five-point scale from 1 (much better) to 5 (much worse). Total Investigator's Assessment Questionnaire scores range from 12 to 60 with lower Investigator's Assessment Questionnaire scores indicating better relative treatment effectiveness.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - ASST degli Spedali Civili di Brescia, Brescia
  - Villa Von Siebenthal, Genzano di Roma
  - Azienda Sanitaria Azienda ospedaliero-universitaria Senese, Siena

REFERENCES:
- [Derived] De Filippis S, Vita A, Cuomo A, Amici E, Giovanetti V, Lombardozzi G, Pardossi S, Altieri L, Cicale A, Dosoli M, Galluzzo A, Invernizzi E, Rodigari P, Mascagni P, Santini C, Falsetto N, Manes MA, Micillo M, Fagiolini A. Treatment satisfaction and effectiveness of Lurasidone on quality of life and functioning in adult patients with schizophrenia in the real-world Italian clinical practice: a prospective 3-month observational study. Ann Gen Psychiatry. 2024 Nov 5;23(1):43. doi: 10.1186/s12991-024-00531-z. PMID 39501351